CLINICAL TRIAL: NCT06327659
Title: Efficacy of Using 50 ml Syringe Manual Thrombectomy Catheter in Patients With Heavy Thrombus Burden Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Efficacy of Using 50 ml Syringe Manual Thrombectomy Catheter in Primary PCI With Heavy Thrombus Burden
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Arafa Gomaa, Cardiology consultant, Helwan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Thrombectomy by 50 ml syringe
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; Thrombosis Cardiac
Keywords: STEMI; heavy thrombus burden; manual thrombectomy; 50 mL syringe
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator)
  Interventions: Device: 30 mL syringe manual thrombectomy catheter
- Group II (Experimental)
  Interventions: Device: 50 mL syringe manual thrombectomy catheter

INTERVENTIONS:
Device: 30 mL syringe manual thrombectomy catheter — 30 mL syringe manual thrombectomy catheter
  Arms: Group I
Device: 50 mL syringe manual thrombectomy catheter — 50 mL syringe manual thrombectomy catheter
  Arms: Group II

SUMMARY:
In high thrombus burden subgroup of Acute STEMI, manual aspiration thrombectomy was associated with reduced cardiovascular death but increased stroke or transient ischemic attack. The role of aspiration thrombectomy is still a matter of active debate. Manual aspiration suffers from decreasing aspiration force as the syringe fills with fluid and requires the operator to exchange syringes during the procedure to maintain suction.

DETAILED DESCRIPTION:
Acute ST-segment elevation myocardial infarction (STEMI) poses a major hazard to human life and health due to its high morbidity and deaths. The frequency of STEMI is increasing. Although dual antiplatelet treatment (DAPT) and primary percutaneous coronary intervention (PPCI) have enhanced survival in STEMI suffers during the last 20 years. Complications after myocardial infarction continue to be a major contributor to high mortality and disability.

Treatment focuses on minimizing infarct size by reopening the occluded artery and restoring myocardial perfusion While PPCI is an established treatment option and can reliably re-establish flow, it can also cause distal embolization, resulting in persistent microvascular obstruction and poor myocardial perfusion. Poor myocardial perfusion after PCI is associated with worse left ventricular functional recovery and increased long-term mortality. By removing thrombotic material, aspiration thrombectomy before PCI may reduce the risk of distal embolization and improve myocardial perfusion. A meta-analysis of large randomized trials comparing aspiration thrombectomy and PCI alone found that routine manual aspiration thrombectomy did not improve clinical outcomes. However, in the high thrombus burden subgroup, manual aspiration thrombectomy was associated with reduced cardiovascular death but increased stroke or transient ischemic attack.

For select cardiac populations, particularly those with high thrombus burden, the role of aspiration thrombectomy is still a matter of active debate. Manual aspiration suffers from decreasing aspiration force as the syringe fills with fluid and requires the operator to exchange syringes during the procedure to maintain suction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with STEMI within 12-24 h of symptom onset in native coronary vessel with heavy thrombus burden (Thrombolysis in Myocardial Infarction [TIMI] thrombus grade 4 or 5 on angiography after the guidewire crossed the target lesion)

Exclusion Criteria:

* Very delayed STEMI presentation.
* STEMI with low thrombus burden.
* STEMI with cardiogenic shock.
* Failed recanalization of culprit vessel.
* Complex coronary anatomy candidates for coronary artery bypass graft.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
TIMI flow grade after PCI | During procedure
  Thrombolysis in Myocardial Infarction (TIMI) flow grades:
  * Grade 0: There is no antegrade flow or perfusion beyond the blockage.
  * Grade 1 indicates that the contrast material was able to flow through the blockage during the cineangiographic recording series without totally obstructing the coronary bed distal to the obstruction.
  * Grade 2: The coronary artery distal to the occlusion is opacified by the contrast material at a much slower pace than in regions unaffected by the prior closure.
  * Grade 3: indicates contrast material is cleared from the affected bed at the same rate as it is cleared from an unaffected bed in the same or opposite artery.
MBG after PCI | During procedure
  Myocardial blush grade (MBG):
  * Grade 0: No myocardial blush or contrast density.
  * Grade 1: Minimal myocardial blush or contrast density.
  * Grade 2: Moderate myocardial blush or contrast density but less than that obtained during angiography of a contralateral or ipsilateral non-infarct-related coronary artery.
  * Grade 3: Normal myocardial blush or contrast density comparable with that obtained during angiography of a contralateral or ipsilateral non-infarct-related coronary artery.

SECONDARY OUTCOMES:
Composite rate of occurrence of MACE | 30 days after PCI
  composite of cardiovascular death, recurrent myocardial infarction, stroke, cardiogenic shock, or new or worsening New York Heart Association class IV heart failure
Rate of cardiovascular death | 30 days after PCI
Rate of recurrent myocardial infarction | 30 days after PCI
Rate of stroke | 30 days after PCI
Rate of cardiogenic shock | 30 days after PCI
Rate of NYHA IV heart failure | 30 days after PCI
  New or worsening New York Heart Association class IV heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Arafa Gomaa, MD, Study Director — Helwan University
Locations (1):
- Badr University Hospital, Badr, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbur MCM, Martinez-Avila MC, Madero AI, Nunez JFG, Dominguez JCG. Acute ST-segment elevation myocardial infarction: to be or not to be? Arch Clin Cases. 2022 Apr 6;9(1):19-23. doi: 10.22551/2022.34.0901.10198. eCollection 2022. PMID 35529096
- [Background] Zalewski J, Nowak K, Furczynska P, Zalewska M. Complicating Acute Myocardial Infarction. Current Status and Unresolved Targets for Subsequent Research. J Clin Med. 2021 Dec 16;10(24):5904. doi: 10.3390/jcm10245904. PMID 34945202
- [Background] Anderson JL, Morrow DA. Acute Myocardial Infarction. N Engl J Med. 2017 May 25;376(21):2053-2064. doi: 10.1056/NEJMra1606915. No abstract available. PMID 28538121
- [Background] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX, Anderson JL, Jacobs AK, Halperin JL, Albert NM, Brindis RG, Creager MA, DeMets D, Guyton RA, Hochman JS, Kovacs RJ, Kushner FG, Ohman EM, Stevenson WG, Yancy CW; American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2013 Jan 29;127(4):e362-425. doi: 10.1161/CIR.0b013e3182742cf6. Epub 2012 Dec 17. No abstract available. PMID 23247304
- [Background] Henriques JP, Zijlstra F, Ottervanger JP, de Boer MJ, van 't Hof AW, Hoorntje JC, Suryapranata H. Incidence and clinical significance of distal embolization during primary angioplasty for acute myocardial infarction. Eur Heart J. 2002 Jul;23(14):1112-7. doi: 10.1053/euhj.2001.3035. PMID 12090749
- [Background] Mathews SJ, Parikh SA, Wu W, Metzger DC, Chambers JW, Ghali MGH, Sumners MJ, Kolski BC, Pinto DS, Dohad S. Sustained Mechanical Aspiration Thrombectomy for High Thrombus Burden Coronary Vessel Occlusion: The Multicenter CHEETAH Study. Circ Cardiovasc Interv. 2023 Feb;16(2):e012433. doi: 10.1161/CIRCINTERVENTIONS.122.012433. Epub 2023 Feb 21. PMID 36802804
- [Background] Jolly SS, Cairns JA, Lavi S, Cantor WJ, Bernat I, Cheema AN, Moreno R, Kedev S, Stankovic G, Rao SV, Meeks B, Chowdhary S, Gao P, Sibbald M, Velianou JL, Mehta SR, Tsang M, Sheth T, Dzavik V; TOTAL Investigators. Thrombus Aspiration in Patients With High Thrombus Burden in the TOTAL Trial. J Am Coll Cardiol. 2018 Oct 2;72(14):1589-1596. doi: 10.1016/j.jacc.2018.07.047. PMID 30261959
- [Background] Kobkitsuksakul C, Jaroenngarmsamer T. Comparison of vacuum pressure syringe aspiration technique with penumbra aspiration thrombectomy system: an in vitro study. Hong Kong J Radiol 2021; 24:47-
- [Background] Weinsaft JW, Kim J, Medicherla CB, Ma CL, Codella NC, Kukar N, Alaref S, Kim RJ, Devereux RB. Echocardiographic Algorithm for Post-Myocardial Infarction LV Thrombus: A Gatekeeper for Thrombus Evaluation by Delayed Enhancement CMR. JACC Cardiovasc Imaging. 2016 May;9(5):505-15. doi: 10.1016/j.jcmg.2015.06.017. Epub 2015 Oct 14. PMID 26476503
- [Background] Lashin H, Olusanya O, Smith A, Bhattacharyya S. Left Ventricular Ejection Fraction Correlation With Stroke Volume as Estimated by Doppler Echocardiography in Cardiogenic Shock: A Retrospective Observational Study. J Cardiothorac Vasc Anesth. 2022 Sep;36(9):3511-3516. doi: 10.1053/j.jvca.2022.05.009. Epub 2022 May 10. PMID 35662515
- [Background] Lee OH, Kim Y, Son NH, Roh JW, Im E, Cho DK, Choi D. Comparison of Distal Radial, Proximal Radial, and Femoral Access in Patients with ST-Elevation Myocardial Infarction. J Clin Med. 2021 Aug 2;10(15):3438. doi: 10.3390/jcm10153438. PMID 34362221
- [Background] Suleiman S, Coughlan JJ, Arockiam S, Arnous S, Kiernan TJ. Pre-Percutaneous Coronary Intervention TIMI Flow Grade in STEMI Patients Treated with Pre-Hospital Ticagrelor Loading. Ir Med J. 2022 Mar 16;115(3):564. PMID 35532897
- [Background] Gibson CM, de Lemos JA, Murphy SA, Marble SJ, McCabe CH, Cannon CP, Antman EM, Braunwald E; TIMI Study Group. Combination therapy with abciximab reduces angiographically evident thrombus in acute myocardial infarction: a TIMI 14 substudy. Circulation. 2001 May 29;103(21):2550-4. doi: 10.1161/01.cir.103.21.2550. PMID 11382722
- [Background] Gibson CM, Cannon CP, Murphy SA, Ryan KA, Mesley R, Marble SJ, McCabe CH, Van De Werf F, Braunwald E. Relationship of TIMI myocardial perfusion grade to mortality after administration of thrombolytic drugs. Circulation. 2000 Jan 18;101(2):125-30. doi: 10.1161/01.cir.101.2.125. PMID 10637197